CLINICAL TRIAL: NCT07210671
Title: Prospective Evaluation of the Treatment of Cancer Associated Superficial Venous
Acronym: SUPERCAT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2024_843_0121
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Superficial Vein Thrombosis; Cancer; Venous Thrombosis
Keywords: Superficial vein thrombosis; cancer; venous thrombosis
MeSH Terms: conditions — Neoplasms; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Superficial venous thrombosis (SVT) is very common in clinical practice. What's more, around 15- 20% of SVTs occur in the context of cancer. Today, cancer patients are excluded from therapeutic trials for DVT. There is therefore no high-level evidence-based treatment recommendation for these patients. Recent data suggest that the course of cancer-associated DVT is similar to that of cancer-associated deep vein thrombosis (DVT). However, there are currently few prospective data on the evolution of cancer-associated DVT in relation to the treatment used. Due to the absence of clear recommendations of treatment in case of SVT associated with cancer the investigators will perform a prospective observational study to evaluate the efficacy of different regiment of anticoagulant treatment ordered in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* Patient affiliated to a social security scheme
* Patient who understands French
* Patient with superficial venous thrombosis of the lower and upper limbs confirmed by a Doppler ultrasound less than one month old.
* Patient with active cancer:
* Cancer treatment within the last 6 months,
* Detectable tumor disease, cancer treatment within the last 6 months, ongoing hormone therapy for cancer, palliative cancer.
* The patient has received potentially non-curative cancer treatment (notably palliative chemotherapy).
* Progression shows that the cancer treatment was not curative (due to recurrence or progression under treatment) (particularly in the case of recurrence after surgery)

Exclusion Criteria:

* Patients under legal protection
* Patients with concomitant pulmonary embolism
* Patient with proximal or distal deep vein thrombosis
* Patient treated with anticoagulant therapy for another indication
* Patient with a contraindication to anticoagulation: Thrombocytopenia less than 30,000 elements/mm3, active bleeding or history of severe bleeding.
* Patient opposed to participation in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with active cancer:
  * Cancer treatment within the last 6 months,
  * Detectable tumor disease, cancer treatment within the last 6 months, ongoing hormone therapy for cancer, palliative cancer.
  * The patient has received potentially non-curative cancer treatment (notably palliative chemotherapy).
  * Progression shows that the cancer treatment was not curative (due to recurrence or progression under treatment) (particularly in the case of recurrence after surgery)
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
risk (in %) of recurrence of VTE | at 3-month follow-up
  risk of recurrence of VTE at 3-month follow-up in patients with cancer-associated SVT.

SECONDARY OUTCOMES:
association (%) between initial treatment and the risk of SVT recurrence | at 3 months
association (%) between initial treatment and the risk of SVT recurrence | at 6 months
association (%) between initial treatment and the risk of SVT recurrence | at 12 months
Association (%) between initial treatment and the occurrence of pulmonary embolism (PE) | at 12 months
Association (%) between initial treatment and the occurrence of pulmonary embolism (PE) | at 3 months
Association (%) between initial treatment and the occurrence of DVT | at 3 months
Association (%) between initial treatment and the occurrence of pulmonary embolism (PE) | at 6 months
Association (%) between initial treatment and the occurrence of DVT | at 12 months
Association (%) between initial treatment and the occurrence of DVT | at 6 months
association (%) between initial treatment and bleeding events | at 6 months
association (%) between initial treatment and bleeding events | at 3 months
association (%) between initial treatment and bleeding events | at 12 months
association(%) between initial treatment and all-cause death | at 3 months
association(%) between initial treatment and all-cause death | at 6 months
association(%) between initial treatment and all-cause death | at 12 months
rates of recurrence of symptomatic vs. incidental VTE | at 3 months
rates of recurrence of symptomatic vs. incidental VTE | at 6 months
rates of recurrence of symptomatic vs. incidental VTE | at 12 months
rate of confirmed cancer in patients with TVS suspected of having cancer. | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No